CLINICAL TRIAL: NCT02120469
Title: Phase I/IB Trial of Eribulin and Everolimus in Patients With Triple Negative Metastatic Breast Cancer
Brief Title: Eribulin Mesylate and Everolimus in Treating Patients With Triple-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14036; NCI-2014-00844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14036 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor-negative; Stage IV Breast Cancer; Triple-negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Everolimus; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (everolimus, eribulin mesylate) (Experimental): Patients receive everolimus PO QD on days 1-21 and eribulin mesylate IV on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Drug: eribulin mesylate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: eribulin mesylate — Given IV
  Other Names: B1939; E7389; ER-086526; halichrondrin B analog
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase I/IB trial studies the side effects and best dose of eribulin mesylate and everolimus in treating patients with breast cancer that does not have estrogen receptors, progesterone receptors, or large amounts of human epidermal growth factor receptor 2 protein (triple-negative) and has spread to other places in the body (metastatic). Eribulin mesylate and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of everolimus and eribulin (eribulin mesylate), and determine the recommended Phase IB dose (RP2D) of the drug combination in patients with resistant metastatic triple negative breast cancer (TNBC). (Phase I) II. To evaluate the event-free survival (EFS) rate for patients with resistant metastatic TNBC at the RP2D of everolimus and eribulin to determine if the drug combination is worthy of further study. (Phase IB)

SECONDARY OBJECTIVES:

I. To determine response rate in patients with resistant metastatic TNBC. (Phase IB) II. To determine overall survival (OS) in patients with resistant metastatic TNBC. (Phase IB) III. To determine toxicity in patients with resistant metastatic TNBC. (Phase IB) IV. To determine pharmacokinetics (PK) for everolimus and eribulin in patients with resistant metastatic TNBC. (Phase IB) V. To collect blood, skin punch biopsies, and tumor biopsies before and after treatment from all patients and perform proteomic analysis to determine the level of inhibition of the phosphatidylinositol 3 kinase (PI3K) pathway in tumor cells versus non-therapeutic targets. (Phase IB)

OUTLINE: This is a dose-escalation study of everolimus.

Patients receive everolimus orally (PO) once daily (QD) on days 1-21 and eribulin mesylate intravenously (IV) on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 21 days and then periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed stage IV TNBC (patients who had metastatic disease within 6 months of lumpectomy or mastectomy for treatment of TNBC may be excused from repeat biopsy)
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion; newly obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1; subjects for whom newly obtained samples cannot be provide (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the study principle investigator (PI)
* Patients must have had prior treatment with anthracyclines and/or taxanes (resistant) or platinum including adjuvant or neoadjuvant therapy
* Both measurable as well as non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, will be allowed
* Patients with chemotherapy for metastatic disease (patients with 0-3 prior lines of chemotherapy for metastatic breast cancer [MBC])
* Life expectancy of >= 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Hemoglobin >= 9.0 g/dl
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 times the upper limit of normal (ULN)
* Total bilirubin less =< to 1 times ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< to 2.5 times the ULN if no liver metastases; for patients with known liver metastases, AST and ALT must be =< to 5 times the ULN
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for up to 8 weeks after ending treatment; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Be willing to use dexamethasone mouthwash as directed

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events (AEs) due to agents administered > 3 weeks prior to entering the study
* Patients may not be receiving any other investigational agents
* Patients with symptomatic brain metastases are excluded from this clinical trial
* Uncontrolled current illness including, but not limited to, ongoing or active infection (> grade 2 based on the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version [v]4.0), symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women
* Prior eribulin use
* Patients with human immunodeficiency virus (HIV), chronic hepatitis B, or chronic hepatitis C (known from the existing medical record)
* Concomitant use with strong or moderate cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)/P-glycoprotein (PgP) inhibitors and CYP3A4/PgP inducers
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after ending treatment; highly effective contraception methods include combination of any two of the following:

  * Use of oral, injected or implanted hormonal methods of contraception or
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Total abstinence
  * Male/female sterilization

Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential

* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Noncompliant with oral medication and/or dexamethasone mouth wash

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yuan, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - South Pasadena Cancer Center, South Pasadena, California

REFERENCES:
- [Derived] Lee JS, Yost SE, Blanchard S, Schmolze D, Yin HH, Pillai R, Robinson K, Tang A, Martinez N, Portnow J, Wen W, Yim JH, Brauer HA, Ren Y, Luu T, Mortimer J, Yuan Y. Phase I clinical trial of the combination of eribulin and everolimus in patients with metastatic triple-negative breast cancer. Breast Cancer Res. 2019 Nov 8;21(1):119. doi: 10.1186/s13058-019-1202-4. PMID 31703728

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level B1: everolimus 5mg; eribulin 1.1mg/m^2; 10 mL dexamethasone mouthwash
  Patients receive 5mg everolimus PO QD on days 1-21 and 1.1 mg/m^2 eribulin mesylate IV on days 1 and 8 and 10 mL of alcohol-free dexamethasone 0.5 mg/5 mL oral solution, swish for 2 min and spit, 4 times daily. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Dose Level A1: everolimus 5mg; eribulin 1.4mg/m^2
  Patients receive 5 mg everolimus PO QD on days 1-21 and 1.4 mg/m^2 eribulin mesylate IV on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Dose Level A2: everolimus 7.5mg; eribulin 1.4mg/m^2
  Patients receive 7.5 mg everolimus PO QD on days 1-21 and 1.4 mg/m^2 eribulin mesylate IV on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level B1 | Dose Level A1 | Dose Level A2
Started | 13 | 10 | 4
Completed | 12 | 10 | 3
Not Completed | 1 | 0 | 1
Not completed — HER-2/neu-amplified | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Level A1: 5mg everolimus; 1.4 mg/m^2 eribulin mesylate
  Patients receive 5mg everolimus PO QD on days 1-21 and 1.4 mg/m^2 eribulin mesylate IV on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Dose Level A2: 7.5mg everolimus; 1.4 mg/m^2 eribulin mesylate
  Patients receive 7.5mg everolimus PO QD on days 1-21 and 1.4 mg/m^2 eribulin mesylate IV on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Dose Level B1 | Dose Level A1 | Dose Level A2 | Total
Number analyzed (Participants) | 13 | 10 | 4 | 27
Age, Continuous [Median (Full Range); unit: years] | 56 [36 to 76] | 52.5 [41 to 68] | 50.5 [45 to 64] | 55 [36 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 4 | 27
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 2 | 9
  Not Hispanic or Latino | 10 | 6 | 2 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 10 | 5 | 3 | 18
  Race: Asian/Pacific Islander | 1 | 1 | 1 | 3
  Race: Black | 1 | 1 | 0 | 2
  Race: Unknown | 1 | 3 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 10 | 4 | 27
ECOG performance status [Count of Participants; unit: Participants]
  Fully active, able to carry on all pre-disease performance without restriction | 4 | 3 | 1 | 8
  Restricted in physically strenuous activity but ambulatory and able to do work of a light nature | 8 | 4 | 3 | 15
  Ambulatory and capable of all selfcare but unable to carry out any work activities | 1 | 3 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicity (DLT) (Phase I) and the Recommended Phase IB Dose (RP2D)
Description: DLT defined as an adverse event (AE) or abnormal laboratory value as at least possibly related to the study medication and meets any of the criteria per NCI CTCAE v4.0.
Time Frame: First cycle on treatment, up to 21 days
Population: Number analyzed for DLT only include participants that are evaluable. A1: 1 participant was not evaluable due to progression prior to completion of first two cycles and 1 participant was not evaluable due to toxicity attributed to diabetes.
  A2: 1 participant was not evaluable due to HER2+ repeat biopsy. B1: 1 participant was not evaluable due to HER2+ repeat biopsy.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level A1: everolimus 5mg; eribulin 1.4mg/m^2
  Patients receive 5mg everolimus PO QD on days 1-21 and 1.4 mg/m^2 eribulin mesylate IV on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Dose Level A2: everolimus 7.5mg; eribulin 1.4mg/m^2
  Patients receive 7.5mg everolimus PO QD on days 1-21 and 1.4 mg/m^2 eribulin mesylate IV on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level B1 | Dose Level A1 | Dose Level A2
Number analyzed (Participants) | 12 | 8 | 3
Participants | 4 | 4 | 2
Statistical Analysis 1: Comparison: Dose Level B1 vs Dose Level A1 vs Dose Level A2; Test type: Other; Dose level B1 (eribulin 1.1 mg/m2 days 1 and 8 every 3 weeks with everolimus 5 mg daily) was defined as the highest dose with acceptable toxicity (RP2D)

2. Primary Outcome: Number of Subjects With Disease Progression Using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (Phase IB)
Description: Progression determined using response evaluation criteria in solid tumors (RECIST) version 1.1 or showed clinical progression. RECIST criteria for progression includes: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started (including the baseline scan if that is the smallest), and at least a 5mm increase or the appearance of new lesions. Rates and associated 95% confidence limits will be estimated.
Time Frame: Up to 2 years
Population: 2 participants (1 on dose level A2 and 1 on dose level B1) were not evaluable for response because they were determined to be HER2+ on repeat biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level B1 | Dose Level A1 | Dose Level A2
Number analyzed (Participants) | 12 | 10 | 3
Participants | 10 | 8 | 3

3. Secondary Outcome: Number of Participants With Grade 3 or Higher Toxicities (Phase IB)
Description: Will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for grade 3 or higher toxicities attributed to eribulin mesylate or everolimus.
Time Frame: On treatment, 21 days per cycle up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level B1 | Dose Level A1 | Dose Level A2
Number analyzed (Participants) | 13 | 10 | 4
Participants | 8 | 5 | 3

4. Secondary Outcome: Best Response Using the RECIST (Phase IB)
Description: RECIST Criteria:
  Complete Response (CR): Disappearance of all target lesions. Lymph node CR is when the lymph node has decreased to less than 10mm in the short axis.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started (including the baseline scan if that is the smallest), and at least a 5mm increase or the appearance of new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level B1 | Dose Level A1 | Dose Level A2
Number analyzed (Participants) | 12 | 10 | 3
Participants
  Partial Remission | 5 | 3 | 1
  Stable Disease | 6 | 2 | 1
  Progressive Disease | 1 | 5 | 1

5. Secondary Outcome: Median Overall Survival (Phase IB)
Description: Kaplan Meier methods will be used to estimate the median and 95% confidence limits across all dose levels per protocol plan.
Time Frame: From start of treatment to death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Everolimus, Eribulin Mesylate)
Number analyzed (Participants) | 25
months | 8.3 [5.5 to NA] — Due to insufficient number of participants with events

6. Secondary Outcome: Median Progression Free Survival (Phase IB)
Description: Kaplan Meier methods will be used to estimate the median and 95% confidence limits over all dose levels per protocol plan.
Time Frame: Form the date treatment begins until the first date on which recurrence, progression, or death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Everolimus, Eribulin Mesylate)
Number analyzed (Participants) | 25
months | 2.6 [2.1 to 4.0]

ADVERSE EVENTS:
Time Frame: While on study, an average of 9 months
Arm/Group | Dose Level B1 | Dose Level A1 | Dose Level A2
All-Cause Mortality (participants affected / at risk) | 6/13 | 10/10 | 3/4
Serious Adverse Events (participants affected / at risk) | 1/13 | 3/10 | 1/4
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level B1 (N=13) | Dose Level A1 (N=10) | Dose Level A2 (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1
Infections and infestations - other (Infections and infestations) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level B1 (N=13) | Dose Level A1 (N=10) | Dose Level A2 (N=4)
Anemia (Blood and lymphatic system disorders) | 10 | 9 | 4
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 4 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 6 | 8 | 2
Tricuspid valve disease (Cardiac disorders) | 2 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 5 | 1
Diarrhea (Gastrointestinal disorders) | 6 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 9 | 5 | 4
Nausea (Gastrointestinal disorders) | 8 | 4 | 2
Oral pain (Gastrointestinal disorders) | 0 | 3 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Death NOS (General disorders) | 1 | 1 | 0
Edema face (General disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 3 | 2
Facial pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 12 | 8 | 2
Fever (General disorders) | 2 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 1
Infusion site extravasation (General disorders) | 1 | 0 | 0
Localized edema (General disorders) | 2 | 1 | 0
Non-cardiac chest pain (General disorders) | 4 | 1 | 0
Pain (General disorders) | 4 | 4 | 0
Gum infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 2 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 2
Alkaline phosphatase increased (Investigations) | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 5 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 0
CD lymphocytes decreased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 6 | 3
Neutrophil count decreased (Investigations) | 11 | 9 | 4
Platelet count decreased (Investigations) | 2 | 5 | 1
Weight loss (Investigations) | 8 | 2 | 2
White blood cell decreased (Investigations) | 10 | 9 | 4
Alkalosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 4 | 7 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 5 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 2
Dysgeusia (Nervous system disorders) | 4 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 6 | 2 | 1
Movements involuntary (Nervous system disorders) | 0 | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1 | 3
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 6 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Spasticity (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 2
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 3 | 2
Personality change (Psychiatric disorders) | 0 | 1 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 2 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 2 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Hot flashes (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 10 | 9 | 2
Hypotension (Vascular disorders) | 5 | 1 | 0
Lymphedema (Vascular disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02120469/Prot_SAP_000.pdf